CLINICAL TRIAL: NCT05060159
Title: A Pilot Randomized Control Trial of Conventional Hemodialysis Versus Post-Dilution Hemofiltration as First Treatment of Renal Replacement Therapy in Chronic Kidney Disease: The DA-VINCI Study
Brief Title: Conventional Hemodialysis Versus Post-Dilution Hemofiltration in Incident RRT
Acronym: DA-VINCI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Magdalena Madero, MD, Instituto Nacional de Cardiologia Ignacio Chavez
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PT-19-121
Record Dates: First submitted 2021-03-31; First posted 2021-09-29 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Dialysis; Complications; Hemodialysis Complication; Cerebral Edema; Cognitive Impairment
Keywords: hemodialysis; hemofiltration; cognitive impairment; post-dialytic syndrome; brain magnetic resonance imaging
MeSH Terms: conditions — Brain Edema; Cognitive Dysfunction | interventions — Hemofiltration

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hemodialysis (No Intervention): Conventional hemodialysis
- Hemofiltration (Experimental): Postdilutional hemofiltration
  Interventions: Other: Hemofiltration

INTERVENTIONS:
Other: Hemofiltration — Postdilutional Hemofiltration
  Arms: Hemofiltration

SUMMARY:
Patients with chronic kidney disease (CKD) with criteria for renal replacement therapy (RRT) including uremic syndrome, have a stable state of hyperosmolarity due to urea despite not being an osmotically inactive ion. Also, these patients have alterations in urea transporters in the central nervous system (CNS) conferring a risk of neurological involvement due to an abrupt decrease in serum urea causing manifestations of the post-dialytic syndrome.

Hemodialysis results in rapid removal of urea from the blood, much faster than the equilibrium rate between the brain and the bloodstream through the blood-brain barrier, resulting in an osmotic gradient that favors movement from water to the brain, causing cerebral edema, intracranial hypertension and dialysis-associated imbalance syndrome. Conventional hemodialysis (HD) uses diffusion and primarily decreases small solutes, while hemofiltration (HF) is based on convection that provides clearance mainly of medium-size molecules and small solutes with a slower rate of reduction.

DETAILED DESCRIPTION:
Currently, there is little information about which is the safest modality in the first session of intermittent hemodialysis. Other than dialysis-associated imbalance syndrome, there is no evidence exploring the neurocognitive effects of the first hemodialysis session. Cognitive impairment is defined as a new deficit in two or more areas of cognitive function and its progression is associated with impaired kidney function. Most of the dysfunctions reported are in the domains of orientation, attention and executive functions. Therefore, the recognition of cognitive impairment can be done with tools such as the Minimental State Examination (MMSE) and the Montreal Cognitive Assessment (MOCA) test. Brain magnetic resonance imaging (MRI) can identify brain lesions such as 'silent' infarcts, microbleeds and white matter abnormalities in patients with CKD with and without RRT. Diffusion-weighted MRI before and after HD has shown brain edema in rats with dialysis-associated imbalance syndrome. In fact, there is evidence from brain MRI that before first HD session patients have interstitial cerebral edema, which worsens after the first HD treatment.

Because there is no clear evidence to support the choice of the modality in the first session and the prescription is still based on personal experiences and shared views. Therefore, we conducted a pilot study to determine the safest hemodialysis modality with the lowest risks and neurocognitive effects for patients with CKD and first HD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age > 17 years
* Both gender
* CKD stage 5 with clinical or biochemical criteria to kidney replacement therapy initiation that includes:
* Urea nitrogen > 80 mg/dl
* Hyperkalemia
* Fluid overload
* Metabolic acidosis (ph < 7.2 and/or bicarbonate <12)

Exclusion Criteria:

* Visual disturbances
* Altered mental status at enrollment
* Hypothyroidism without optimal supplementation
* Advanced neoplasia
* Acute kidney injury

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2021-03-06 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Neurological status | Immediately after intervention
  Before and after the intervention, the Minimental State Examination (MMSE) and Montreal Cognitive Assessment (MOCA) test were applied in all patients as well as brain magnetic resonance imaging (MRI) was performed in 7 patients from conventional HD group and 8 patients from post-dilution HF group before and after the intervention.
  We used both neurocognitive test and MRI to determine the safest HD modality (conventional hemodialysis versus hemofiltration) with the lowest neurological risks and neurocognitive effects for patients with CKD and incident RRT.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Nacional de Cardiología Dr. Ignacio Chávez, Mexico City, México City, Mexico

REFERENCES:
- [Derived] Kulkarni M, Prabhu AR, Rao IR, Nagaraju SP. Interventions for preventing haemodialysis dysequilibrium syndrome. Cochrane Database Syst Rev. 2024 May 22;5(5):CD015526. doi: 10.1002/14651858.CD015526.pub2. PMID 38775299
- [Derived] Jimenez EV, Nunez GC, Lerma A, Lerma C, Gonzalez AM, Perez-Grovas H, Gil SL, Madero M. Neurocognitive Function with Conventional Hemodialysis versus Post-Dilution Hemofiltration as Initial Treatment in ESKD Patients: A Randomized Controlled Trial - The DA-VINCI Study. Blood Purif. 2024;53(2):130-137. doi: 10.1159/000534823. Epub 2023 Oct 27. PMID 37899042